CLINICAL TRIAL: NCT07321730
Title: Surgeons' Ability to Predict Pathological and Molecular Features of Peritoneal Carcinomatosis in Ovarian Cancer
Acronym: Visual-PC
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 8151
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: VISUAL PC - SURVEY 2.0 — Survey for surgeons in order to study their ability to recognize macroscopic features for selecting appropriate treatment strategies in patients with abdominal malignancies.

SUMMARY:
Epithelial ovarian cancer (EOC) presents with peritoneal carcinomatosis (PC) at diagnosis in approximately two-thirds of cases. Diagnostic laparoscopy is pivotal to assess disease extent and to guide the choice between primary cytoreductive surgery (PCS) and neoadjuvant chemotherapy followed by interval cytoreductive surgery (ICS). The Predictive Index Value (PIV) provides a quantitative estimate of resectability, but it does not systematically capture qualitative intraoperative descriptors. Growing evidence suggests that macroscopic features (e.g., nodularity, plaques, omental cake, infiltrative vs expansile growth, margin definition, vascularization, and tissue retraction) may correlate with histotype and molecular profile, and possibly with chemosensitivity. However, surgeons' ability to recognize these visual patterns in a standardized manner has not been systematically investigated.

This cross-sectional survey will assess whether gynecologic oncologic surgeons managing PC can: distinguish malignant metastases from benign tumor-like lesions; associate morphologic patterns with tumor histotypes (type I vs type II EOC and ovarian metastases from other primaries); classify high-grade serous ovarian cancer (HGSOC) growth pattern as infiltrative vs exophytic/expansile; and infer molecular status from macroscopic appearance. The secondary objective is to compare accuracy and confidence between senior and junior surgeons.

Seventy to eighty surgeons will complete an online survey (Microsoft Forms) presenting anonymized laparoscopic images retrospectively selected from routinely recorded diagnostic-laparoscopy videos of 19 consented patients with advanced EOC and PC. Participants will classify each case using predefined categories and rate confidence on a 5-point Likert scale. Analyses will be primarily descriptive (counts/percentages); senior vs junior comparisons will use χ²/Fisher's exact tests for categorical variables and the Mann-Whitney U test for ordinal measures, as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Gynecologic oncologists involved in the surgical management of ovarian cancer
* Gynecology oncology surgeons with a high level of expertise in OC surgery, with years of independent surgical practice
* Gynecology oncology surgeons holding a leading/responsible position.
* Gynecology oncology surgeons in training in oncologic surgery for ovarian cancer.
* Gynecology oncology surgeons with few years of experience in oncologic surgery for ovarian cancer.
* Patients with advanced OC who underwent diagnostic laparoscopy, with the intra- operative video available as part of routine clinical practice.
* The patient's written informed consent will be required to authorize the use of images extracted from diagnostic laparoscopy videos.
* The informed consent of the participating gynecologic oncologists will be collected electronically through the survey (e.g., via checkbox or digital acceptance).

Exclusion Criteria:

* Surgeons not involved in the surgical management of ovarian cancer.
* Incomplete questionnaires or questionnaires not completed according to the provided instructions

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gynecologic oncologists with surgical experience in the management of ovarian cancer, both senior and young surgeons. A senior surgeon is a reference surgeon with a high level of expertise in ovarian cancer (OC) surgery, typically with years of independent surgical practice or holding a leadership or responsible role. The junior surgeon is a surgeon in advanced training or with a few years of experience in complex oncologic surgery for ovarian cancer.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Visual pattern of ovarian cancer | 1 month
  To assess the ability of gynecologic oncologic surgeons to visually recognize pathological and molecular features of peritoneal carcinomatosis in advanced ovarian cancer.

SECONDARY OUTCOMES:
Differences beetween senior and junior surgeons | 1 month
  To compare diagnostic accuracy between senior and junior surgeons.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Fagotti, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS